CLINICAL TRIAL: NCT00477503
Title: Phase 1 Study Nuclear Imaging of Human CSF Flow Using Ga-67 Citrate and In-111 DTPA
Brief Title: Nuclear Imaging of Human CSF Flow Using Ga-67 Citrate and In-111 DTPA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: One participant enrolled, study terminated .
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0623
Record Dates: First submitted 2007-05-21; First posted 2007-05-23 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Central Nervous System Tumors; Brain Tumors
Keywords: Central Nervous System Tumors; Brain Tumors; Leptomeningeal Metastasis; Cerebral Spinal Fluid; Human CSF Flow; Nuclear Imaging; Gallium-67 Citrate; In-111 DTPA
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Meningeal Carcinomatosis | interventions — gallium citrate; Gallium-67; Pentetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): Ga-67 citrate injection alone for individuals with cancer cells in cerebral spinal fluid (CSF), no earlier treatment for disease.
  Interventions: Drug: Gallium-67 Citrate (Ga-67)
- Group B (Active Comparator): Ga-67 + In 111 DTPA injection for individuals who have cancer cells in CSF, no earlier treatment for disease.
  Interventions: Drug: Gallium-67 Citrate (Ga-67); Drug: In-111 DTPA (In-111 pentetate)
- Group C (Active Comparator): Individuals with tumors in the CSF that have been treated and are now cleared from the CSF, receive standard follow-up care (baseline injection of Ga-67 citrate and In-111 DTPA).
  Interventions: Drug: Gallium-67 Citrate (Ga-67); Drug: In-111 DTPA (In-111 pentetate)

INTERVENTIONS:
Drug: Gallium-67 Citrate (Ga-67) — Group A: Ga-67 citrate injection alone, in the baseline study.
  Group B: Ga-67 and In 111 DTPA injection in the baseline study.
  Group C: Standard of care with Ga-67 and In 111 DTPA injection in baseline study.
Drug: In-111 DTPA (In-111 pentetate) — Group B: Ga-67 and In 111 DTPA injection in the baseline study.
  Group C: Standard of care with Ga-67 and In 111 DTPA injection in baseline study.
  Other Names: DTPA
  Arms: Group B; Group C

SUMMARY:
* Primary Objective will be to evaluate the use of Ga-67 citrate as an alternative radiopharmaceutical for CSF imaging.
* Secondary Objective will be to evaluate the biodistribution, pharmacokinetics and radiation dosimetry of In 111 DTPA and gallium-67 after intrathecal injection during remission of leptomeningeal metastasis (LM) and during LM occurrence, remission and recurrence.

DETAILED DESCRIPTION:
In-111 DTPA is a radioactive dye that is standardly used to check the flow of CSF. Ga-67 citrate has been used to detect inflammation and tumors in other parts of the body, and researchers want to learn if it is also able to detect tumors in the brain and spinal cord.

Before you can be enrolled in this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Blood (about 1-2 tablespoons) will be drawn for routine tests. This routine blood draw will include a pregnancy test for women who are able to have children. To be eligible to take part in this study, the pregnancy test must be negative.

If you are found to be eligible to take part in this study, you will be assigned to 1 of 3 groups. The group you are assigned to will depend on whether tumor cells were found in the CSF during your last spinal fluid exam. If you were found to have cancer cells in the CSF and you have had no earlier treatment for this type of disease, the first 5 participants will be assigned to Group A and will be given Ga-67 citrate injection alone, in the baseline study. The next 5 participants who have cancer cells in the CSF and have had no earlier treatment will be assigned to Group B. Group B will have Ga-67 and In 111 DTPA injection in the baseline study. Otherwise, if the tumors in the CSF have been treated and are now cleared from the CSF, you will be assigned to Group C and will receive standard follow-up care.

At the beginning of the study, you will have an imaging session. This first imaging session is called the "baseline" session. For the imaging, you will lie on a gamma camera table. Depending on which group you are in, one or both of the radioactive dyes will be injected into your CSF through the Ommaya reservoir. If you are in Group B or C, both In-111 DTPA and Ga-67 citrate will be injected over about 2-4 minutes, total. If you are in Group A, Ga-67 citrate alone will be injected over about 2 minutes.

For participants who are 2-17 years old, the doses of In-111 DTPA and Ga-67 citrate will be adjusted to the surface area of your body (a measurement of your body size).

During the hour immediately following the injections, your head, neck, and back areas will be imaged (scanned) in order to see how the CSF flows. After that, you will have scans of your entire body performed in order to see how quickly the radioactive dyes leave from different parts of your body. These whole-body scans will each last 20 minutes. These scans (1 each time) will occur at 1-2, 3-4, 6-8, 22-24, 28-32, 48, and 72 hours after the injections. You will have blood samples collected before injection and during each imaging session in order to measure how much radiation is absorbed by different parts of your brain, spine, and other organs. These blood samples (less than ¼ teaspoon each time) will be drawn during each of the whole-body scans.

If you are in Group A or B, you will receive standard follow-up care for up to 52 weeks after the baseline imaging session. This is in order to check the status of the disease. If the cancer goes into remission (no tumor cells are found in CSF) at any time during the 52 weeks, you will have a follow-up imaging session. The follow-up imaging session will include the same procedures, and In-111 DTPA and/or Ga-67 citrate injections as the baseline imaging session.

If you are in Group C, you will receive standard follow-up care for up to 52 weeks after the baseline imaging session. If the cancer reappears at any time during the 52 weeks, you will have a follow-up imaging session. The follow-up imaging session will include the same procedures, and In-111 DTPA and Ga-67 citrate injections as the baseline imaging session.

Whether you are in Group A, B or C, after your last follow-up imaging session, your participation in this study will be over. If your cancer clears from the spinal fluid, the records from your routine visit to the neuro-oncology clinic will be reviewed to follow your progress until 30 days after the radioisotope injection for your last imaging session. Researchers will review your medical records for potential side effects. If you do not have a clinical visit within a week from that 30th day, the study chair will contact you by phone concerning these matters.

This is an investigational study. In-111 DTPA is commercially available and FDA approved for injection into the CSF. Although Ga-67 citrate is FDA approved for injection into a vein, it is not FDA approved for injection into the CSF. It is commercially available, but injecting it into the CSF has only been authorized for use in research. Up to 20 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have provided informed consent.
* Participants must be 2 years of age or older.
* Participants must have known history of LM as established by CSF cytology.
* Participants must have an Ommaya reservoir implanted at least 2 days before the study.
* Participants with ventriculoperitoneal shunts are eligible as long as the shunt is not in the "open" position during the imaging session.
* Participants with adequate renal and hepatic function. Creatinine =< 1.4 mg/dL Bilirubin =< 2.0 mg/dL BUN =< 30 SGOT (AST), alkaline phosphatase =<3 x upper norm (Institutional norm of SGOT = 7-56 mIU/ml and alkaline phosphatase = 38-126 IU/L.).
* Urine analysis within normal limits.
* Women of child bearing potential (WOCBP) must have a negative serum B-HCG pregnancy test within 7 days of treatment. WOCBP is defined as not post-menopausal for 12 months or no previous surgical sterilization.

Exclusion Criteria:

* Participants on concurrent external beam radiation therapy to the brain or spine during the planned nuclear imaging sessions.
* Participants on concurrent intrathecal chemotherapy during imaging sessions.
* Participants with Karnofsky Performance Scale <50 or Zubrod Performance Scale >2.
* Participants with known or suspected renal or hepatic disease that have not been adequately treated to achieve normalized liver function tests or renal function tests to the above eligible criteria.
* Participants with known history of claustrophobia, as established by medical records or claimed by patient.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To compare Ga-67 citrate with a standard radioactive dye in order to learn if Ga-67 citrate can help doctors to check the flow of CSF for any blockage. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Franklin C Wong, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org